CLINICAL TRIAL: NCT06667388
Title: Effect of Backward Walking Training Versus Forward Walking Training Program to Improve Balance and Mobility in Children With Cerebral Palsy
Brief Title: Effect of Backward Walking Training vs Forward Walking Training to Improve Balance and Mobility in Children With CP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/746
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Chromosomes, Human, 1-3

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Diagnostic Test: Group A
- Group B (Active Comparator)
  Interventions: Combination Product: Grojup B

INTERVENTIONS:
Diagnostic Test: Group A — each participant of this groups will receive 4 weeks of FWT and 4 weeks of BWT (the training order of A group will FWT and BWT), with a washout period of 2 weeks during the post-intervention phase of the 1st period and the pre-intervention phase for the 2nd period.
  Arms: Group A
Combination Product: Grojup B — each participant of B group will receive 4 weeks of BWT and 4 weeks of FWT (the training order of group B will be BWT and FWT, opposite to group A), with a washout period of 2 weeks during the post-intervention phase of the 1st period and the pre-intervention phase for the 2nd period.
  Arms: Group B

SUMMARY:
Children with cerebral palsy frequently experience balance issues and gait impairments; gait training is a crucial component of their rehabilitation because it greatly enhances the children's socialisation and quality of life.

DETAILED DESCRIPTION:
Since there is no known cure for cerebral palsy, the focus of treatment is shifting to enhancing activities like walking and self-care. Enabling the child with cerebral palsy is the ultimate goal of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Only CP patients will be included.
* Patient will be included from Bahawalpur only.
* Patient will be included having minimum age of 10 year.

Exclusion Criteria:

* Other cities patient will not be included.
* Patient less than 10 years age.
* Patient suffering from other neurological conditions.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Pediatric Functional Independent Measure for Children (WeeFIM) | 12 Months
  The Independence Measure for Children (WeeFIM®) is frequently used as a multiple tool in pediatric clinics to assess the self-care, mobility, and psychological well-being of many groups of children, including those with developmental or developmental disabilities.
  The Functional Independence Measure for Children (WeeFIM) is an 18-item, seven-level ordinal scale instrument used to assess a child's typical and consistent performance.Children 0 to <3 years no WeeFIM (or FIM) is required. Children 3 to <12

CONTACTS AND LOCATIONS:
Locations (1):
- sadiq abbasi hospital bwp Contact: jangi wala road BWP, Chak Four Hundred Fifty-four, Pakistan

IPD SHARING:
Plan to Share IPD: No